CLINICAL TRIAL: NCT01835834
Title: Clinical Study on Zirconia Bridges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Prof. Marco Ferrari, Professor, University of Siena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-159
Record Dates: First submitted 2013-04-05; First posted 2013-04-19 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Missing Teeth
Keywords: zirconia crown
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- zirconia bridge restoration (Experimental): The device is a ceramic core made of shaded zirconium with an anatomic contour core with a minimum of 0.6 mm** thickness and minimal connector size of 4.0 x 3.0 / 9.4 (height x width [mm] / area [mm2])** of high strength zirconia framework providing homogenous veneering material thickness as an external coating with 1.0 - 2.0 mm* wall thickness. The core is veneered with dental porcelain at the dental laboratory.
  Intended use and indications:
  NobelProceraTM Bridge Shaded Zirconia consists of an individualized, supporting substructure in a ceramic bridge construction for tooth/teeth replacement.
  NobelProceraTM Bridge Zirconia is intended for patients in need of prosthetic oral reconstruction in order to restore chewing function. Zirconia bridges for natural tooth restorations are customized, designed, and milled from pre-sintered blanks of zirconia. The multi-unit restorations can be placed in all positions in the mouth.
  Interventions: Procedure: zirconia bridge restoration

INTERVENTIONS:
Procedure: zirconia bridge restoration

SUMMARY:
To evaluate the clinical performance and survival rate of NobelProceraTM Bridge Shaded Zirconia on natural teeth in the posterior region for a period of 5 years. The working hypothesis of this clinical study is that industrial centrally produced 3- or 4-unit bridges of shaded yttrium-oxide partially-stabilized (Y-TZP) zirconia (NobelProceraTM Shaded Zirconia) in combination with a veneering ceramic material will show sufficient CDA ratings (80% R+S) and a sufficient survival rate (93%) after 5 years in comparison with a reference level of 95%.

ELIGIBILITY:
Inclusion Criteria:

The subject must be at least 18 (or age of consent), and less than 70 at the time of inclusion.

* The subject is healthy and compliant with good oral hygiene
* The subject is in need of a posterior fixed partial denture restoration of up to 4 units distal of the canines in the maxilla or mandible.
* The subject shall have a stable occlusal relationship with a fully restored, fixed opposing dentition.
* Obtained informed consent from the subject the subject should be available for the 5-year term of the investigation.
* No apical disorder or inflammation of abutment teeth, adjacent and opposing teeth.
* Good gingival / periodontal / periapical status of restoring, opposing and adjacent teeth. Healed situation of soft tissue augmentation is allowed.
* The subject should be available for the 5-year term of the investigation.

Exclusion Criteria:

* The subject is not able to give her/his informed consent to participate.
* Alcohol or drug abuse as noted in patient records or in patient history.
* Reason to believe that the treatment might have a negative effect on the patient's total situation (psychiatric problems), as noted in patient records or in patient history.
* An existing condition where acceptable retention of the restoration is impossible to attain
* Mobility of the tooth to be restored.
* Pathologic pocket formation of 4 mm or greater around the tooth to be restored
* Severe bruxism or other destructive habits
* Amount of attached soft tissue is insufficient (no attached gingiva on the buccal side of the tooth).
* Health conditions, which do not permit the restorative procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
survival rate of NobelProcera™ Bridge Shaded Zirconia | 5 years
  Success and Failure Criteria The CDA index will be used for the success criteria in this investigation. Please see also the criteria in the "clinical parameter" part of this protocol.
  The success and failure criteria to be used in this investigation have been determined as follows:
  A successful NobelProcera™ Bridge Shaded Zirconia is when:
  the CDA index is Romeo or Sierra at delivery and remains so during the study period.
  A surviving NobelProcera™ Bridge Shaded Zirconia is when:
  the restoration is in occlusion and in function, even though all the success criteria are not fulfilled, but is to be regarded as correctable.
  A failed NobelProcera™ Bridge Shaded Zirconia is when:
  the restoration has 1) been removed, 2) fractured, or 3) cannot be classified as a surviving or a successful restoration.